CLINICAL TRIAL: NCT01643525
Title: A NonRandomized, Multicenter, NonSig Risk Study With a NonInv, Passive PressureWave Method of Diagnosing Cerebral Anomalies to Develop a Diag. Algorithm for Cerebral Isch and to Test Sens./Spec. of This Algorithm in Determining Isch Stroke
Brief Title: Study to Test Sensitivity and Specificity of Passive Wave Pressure Device in Determining Ischemic Stroke
Status: Terminated | Type: Observational
Why Stopped: Insufficient Subject Recruitment
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NA_00069985
Record Dates: First submitted 2012-06-29; First posted 2012-07-18 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with Stroke Symptoms: Suspected stroke subjects that present to hospital with stroke symptoms and are evaluated for stroke
  Interventions: Device: Nautilus NeuroWaveTM System
- Normal Cohort: Subjects that are not being evaluated for stroke and are confirmed to have no cerebrovascular disease
  Interventions: Device: Nautilus NeuroWaveTM System

INTERVENTIONS:
Device: Nautilus NeuroWaveTM System — Non-invasive device designed to detect pressure signals from the skull to aid in the diagnosis of ischemic stroke.

SUMMARY:
That the Jan Medical Nautilus NeuroWaveTM system provides significantly higher sensitivity to hyper acute ischemic stroke than does CT.

DETAILED DESCRIPTION:
In spite of the fact that approximately 800,000 strokes are diagnosed in the United States each year, many physicians and patients have approached the management of stroke with a sense of futility. However, within the past 2 decades, following the advent of computerized tomography (CT), medical interest has turned toward stroke and effective interventions to treat and prevent it have received attention.

CT and/or magnetic resonance imaging (MRI) are the typical diagnostic tools used in the event of a stroke alert. These studies are done on an emergent or urgent basis, since, to be effective, treatments for ischemic and hemorrhagic stroke must be delivered soon after onset of the illness. In an effort to institute an appropriate therapeutic regime, laboratory and structural diagnostic studies are required to be done as rapidly as possible to determine pathological etiology, size, and location of concern.

The speed at which a diagnosis is made and a treatment plan established often determines patient outcome and any associated complications. This is especially true when evaluating patients for ischemic stroke where there is a narrow 3 hour window of opportunity in which to resolve the clot with IV .before permanent neurological impairment results, and up to 8 additional hours with the use if intra arterial (IA) t-PA or interventional mechanical embolectomy procedures are utilized. Current treatment modalities include pharmacologic thrombolytic drugs utilized to disrupt or dissolve clots located in the distal vasculature or mechanical intervention in larger vessels. Since many patients do not recognize the symptoms of stroke they do not seek medical attention immediately. Significant time is then often lost from the onset of the stroke before seeking medical help / treatment.

Although the current technologies are quite adequate as diagnostic tools for hemorrhagic stroke and for identifying subdural hematomas, and other pooled blood abnormalities which would preclude t-PA therapy, they are largely ineffective at positively identifying stroke during the limited therapeutic window of time. Positive identification of ischemia itself is rarely possible or practical with CT or within the limited therapeutic window. As such the diagnostic determination and associated treatment decisions are based on the unsatisfactory basis of exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with stroke with known onset < 12 hours prior to enrollment and planned recording with the Nautilus NeuroWave System
* Suspected pathology of following vessels: internal carotid artery, ACA, MCA, PCA, basilar or other anterior or posterior cerebral vessels or normal anatomy
* Subject is planned to undergo standard stroke triage imaging protocol
* Able to understand and provide signed informed consent, or have a Legally Authorized Representative willing to provide informed consent on subject's behalf

Exclusion Criteria:

* Known to meet hospital criteria for brain death
* Not a candidate for CT, MRI
* unknown time of stroke symptom onset.
* Psychologically unstable and not able to cooperate
* Not suitable for participation in this study in the opinion of the Investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with stroke symptoms that are being evaluated for stroke or healthy subjects that have no cerebrovascular disease and are not being evaluated for symptoms of stroke.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nyquist, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Nautilus NeuroWave Recording Arm: Nautilus NeuroWaveTM System
  Nautilus NeuroWaveTM System: Non-invasive device designed to detect pressure signals from the skull to aid in the diagnosis of ischemic stroke.
Period: Overall Study
Arm/Group | Nautilus NeuroWave Recording Arm
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This number reflects all subjects enrolled in study and is not different from the assignment in the Participant Flow.
Arm/Group | Nautilus NeuroWave Recording Arm
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (16.2)
Sex/Gender, Customized [Number; unit: participants]
  Females Known | 16
  Males Known | 7
  Gender Unknown | 6
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Related Adverse Events
Description: Count the number of participants with device related adverse events
Time Frame: 2-3 days, at subject exit (variation of subject exit date depended on when subject obtained their radiology imaging to confirm ischemic stroke)
Measure: Count of Participants; unit: Participants
Arm/Group | Nautilus NeuroWave Recording Arm
Number analyzed (Participants) | 29
Participants | 0

ADVERSE EVENTS:
Time Frame: 2-3 days, at subject exit (variation of subject exit date depended on when subject obtained their radiology imaging to confirm ischemic stroke)
Arm/Group | Nautilus NeuroWave Recording Arm
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No